CLINICAL TRIAL: NCT05435482
Title: Facilitating COVID-19 At-Home Collection Testing Among Korean American Families Through Korean Schools in Northern California
Brief Title: Facilitating COVID-19 Test for Korean Americans Through Korean Schools in Northern California
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of California, San Francisco (Other)
Collaborators: Duke Clinical Research Institute (Other); National Institute on Minority Health and Health Disparities (NIMHD) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: R0102; U24MD016258 (NIH)
Record Dates: First submitted 2022-06-24; First posted 2022-06-28 (Actual); Results first posted 2024-11-15 (Actual); Last update posted 2024-12-11 (Actual); Status verified 2024-11

CONDITIONS: Educational Activities
MeSH Terms: interventions — Educational Status

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- LHE-led (Experimental): Participants will receive 1) LHE outreach/support (2 small group educational sessions via Zoom and 2 individual follow-up calls), 2) COVID-19 at-home antigen test kits, and 3) a written and a video guide to using a test kit
  Interventions: Behavioral: Education; Other: COVID-19 testing kits; Other: Instruction
- Instruction only (Active Comparator): Participants will receive 1) COVID-19 at-home antigen test kits and 2) a written and a video guide to using a test kit
  Interventions: Other: COVID-19 testing kits; Other: Instruction

INTERVENTIONS:
Behavioral: Education — Participants will receive two small group meetings and two follow-up calls
  Arms: LHE-led
Other: COVID-19 testing kits — Participants will receive two COVID-19 at-home antigen test kits.
Other: Instruction — Participants will receive a written guide and a video clip guide to the test kit.

SUMMARY:
In collaboration with Korean Schools of Northern California, the investigators will test if a community-based intervention delivered by lay health educators (LHEs) increases testing uptake among Korean Americans. A pilot cluster randomized controlled trial (RCT) with 300 participants from about 12 Korean Schools will be conducted to evaluate the efficacy of the LHE-led intervention in promoting COVID-19 testing. Participating schools will recruit Korean Schoolteachers as LHEs. According to the group assignment of schools where participants are recruited, the LHE group participants will receive 1) LHE outreach/support, 2) COVID-19 at-home antigen test kits, and 3) the instruction to use the kit while the control group participants will receive test kits and the instruction. Participants will complete an online survey at baseline, weeks 4, and 8. The primary outcome is the COVID-19 testing receipt. The secondary outcomes are intention to get tested, perceived accuracy, benefits and risks of testing, perceived barriers to testing, understanding of negative or positive results, and family members' testing receipt.

DETAILED DESCRIPTION:
Lay Health Educators (LHEs) Korean Schools in Northern California will be classified into two strata by geographic location (urban, suburban/rural). Collaborating with the KSNC, our research team will recruit about 12 schools (6 urban and 6 suburban/rural). Within each stratum, schools will be randomly assigned in a 1-to-1 ratio to either the LHE-plus-instruction condition (LHE condition) or the instruction-only condition (control condition). Participating schools will recruit two teachers as LHEs (LHE condition only), ii) announce the proposed study to enrolled students' parents, iii) recruit KAs from the school and/or community, and iv) distribute at-home antigen test kits to participants. Research staff will contact potential LHEs to conduct a brief telephone screening to find out their eligibility. If they meet the eligibility and provide an informed consent form via DocuSign, they will be invited to attend two training sessions (6 hours, orientation and intervention delivery) over Zoom. During the training sessions, our research team will provide LHEs Orientation Training Manual, which contains background information, project objectives, project description, lay health educator's responsibilities/activities, compensation/assistance, RCT participant's responsibilities/rights/activities, frequently asked questions, and handling challenging situations. LHEs will also receive the instruction to contact the research team if they do not know how to address the problems. The research team will ask LHEs to respect the privacy of others by keeping confidential any information they learn about others during meetings and calls.

RCT participants All individuals recruited by the schools will receive an email from the research team that includes the consent information of the study and a link to the online baseline survey. They may choose to participate by themselves (individually) or participate with a family member who meets the eligibility criteria to participate together. Each school will recruit about 25 individuals. Those who complete the baseline survey will be assigned to LHE condition or control condition, depending on the group assignment of schools where they are recruited. Within the two weeks after each participant completes the baseline survey, a COVID-19 antigen test kit, which FDA authorizes under a EUA, will be provided to each participant. LHE participants will receive 1) LHE outreach/support (2 small group educational sessions via Zoom and 2 individual follow-up calls), 2) short video clips via email on the project overview and the guide to using a test kit (created by the research team in Korean and English), and 3) test kits with written instructions on COVID-19 testing by Centers for Disease Control and Prevention (CDC) in English and Korean. LHE outreach small group educational session is about 1 hour with 2 to 6 people. LHE will present COVID-19 testing and related information (including vaccination and safety practices). Participants in a dyad (self-selected participation mode) will attend the educational sessions together. At these educational sessions, LHE will provide education using PowerPoint presentations with easy-to-understand messages using culturally appropriate images and simple texts to present current information on 1) COVID-19 testing; 2) relevance or reasons for getting tested; 3) the current guidelines for testing/ who should be tested; 4) types of tests available (e.g., PCR, antigens, and antibodies tests in forms of nose swap and saliva tests); 5) understanding test results (positive versus negative) and the limitation of such tests (false negative); 6) the importance of repeated testing, discussing and addressing barriers for testing. LHE may assist in helping the participant use a COVID-19 at-home antigen test kit, including demonstrating the use of the test kit. Participants will be assessed via online survey or by telephone of their choice at baseline, weeks 4 and 8. Participants will receive up to $70 gift cards for completing all the surveys: $20 for baseline, $20 for week 4, and $30 for week 8. Control participants will receive the same components of the LHE condition except for LHE outreach/support. All control participants will be assessed at the same schedule: baseline, weeks 4 and 8. They will receive the same incentives ($70 gift cards for completing all assessments).

ELIGIBILITY:
Inclusion Criteria:

For Lay Health Educators (LHE), inclusion criteria are:

* age 18 and older;
* self-identify as Korean or Korean American;
* fluent in spoken and written Korean; and
* live in communities where participating schools are located.

For RCT participants, inclusion criteria are:

* age 18 and older;
* self-identify as Korean or Korean American;
* read and speak English or Korean;
* live in communities where participating schools are located; and
* have access to a phone to receive follow-up calls from LHEs.

Exclusion Criteria:

• Participating as community advisory group member for the study

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 259 (Actual)
Dates: Start 2022-10-03 (Actual); Primary Completion 2023-04-30 (Actual); Study Completion 2023-06-30 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: JiWon Choi, PhD, Principal Investigator — University of California, San Francisco
Locations (1):
- University of California, San Francisco, San Francisco, California, United States

IPD SHARING:
Plan to Share IPD: Yes
De-identified data will be shared upon request and data use agreement must be signed
Supporting Information: ICF
Time Frame: Approximately 9 months after data completion
Access Criteria: De-identified data will be shared upon request with a data use agreement

RESULTS

PARTICIPANT FLOW:
Recruitment Details: A total of 259 people were recruited. However, 18 clusters were randomized and a total of 220 completed the baseline survey.
Groups:
- LHE-led: Participants recruited by teachers or online platforms completed the initial online survey. Those who met the eligibility and wanted to participate in the project signed the online consent form and completed the baseline online survey. Once at least 10 participants from specific regions (San Francisco/San Mateo, East Bay, Santa Clara, and Sacramento) were gathered through teachers and/or online platforms to form clusters, our research team randomly assigned these clusters to either the intervention or control group.
  Participants received 1) LHE outreach/support (2 small group educational sessions via Zoom and 2 individual follow-up calls), 2) COVID-19 at-home antigen test kits, and 3) a written and a video guide to using a test kit
- Instruction Only: Participants recruited by teachers or online platforms completed the initial online survey. Those who met the eligibility and wanted to participate in the project signed the online consent form and completed the baseline online survey. Once at least 10 participants from specific regions (San Francisco/San Mateo, East Bay, Santa Clara, and Sacramento) were gathered through teachers and/or online platforms to form clusters, our research team randomly assigned these clusters to either the intervention or control group.
  Participants received 1) COVID-19 at-home antigen test kits and 2) a written and a video guide to using a test kit.
Period: Overall Study
Arm/Group | LHE-led | Instruction Only
Started | 109 | 111
Completed | 102 | 106
Not Completed | 7 | 5

BASELINE CHARACTERISTICS:
Groups:
- Instruction Only: Participants received 1) COVID-19 at-home antigen test kits and 2) a written and a video guide to using a test kit.
- LHE-led: Participants received 1) LHE outreach/support (2 small group educational sessions via Zoom and 2 individual follow-up calls), 2) COVID-19 at-home antigen test kits, and 3) a written and a video guide to using a test kit
- Total: Total of all reporting groups
Arm/Group | Instruction Only | LHE-led | Total
Number analyzed (Participants) | 111 | 109 | 220
Age, Continuous [Mean (Standard Deviation); unit: years] | 44.2 (11.4) | 42.8 (11.6) | 43.5 (11.5)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 75 | 85 | 160
  Male | 36 | 24 | 60
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  Korean | 111 | 109 | 220
Region of Enrollment [Number; unit: participants]
  United States | 111 | 109 | 220
Intention to get tested for COVID-19 as needed [Count of Participants; unit: Participants] | 65 | 66 | 131
COVID-19 Testing receipts in the past 30 days [Count of Participants; unit: Participants] | 22 | 29 | 51

OUTCOME MEASURES:

1. Primary Outcome: Proportion of Participants Who Has Been Tested for COVID-19 During the Study Period
Description: Participants are asked to self-report whether they have been tested for COVID-19 since participation of the intervention program
Time Frame: Week 4
Measure: Count of Participants; unit: Participants
Arm/Group | Instruction Only | LHE-led
Number analyzed (Participants) | 109 | 104
Participants | 34 | 51

2. Primary Outcome: Proportion of Participants Who Has Been Tested for COVID-19 During the Study
Description: as for outcome 1
Time Frame: Week 8
Measure: Count of Participants; unit: Participants
Arm/Group | Instruction Only | LHE-led
Number analyzed (Participants) | 105 | 102
Participants | 30 | 28

3. Secondary Outcome: Intention to Get Tested for COVID-19
Description: Participants are asked to rate their Intention to get tested for COVID-19. A score at 3 or higher is considered as having intention to get tested for COVID-19
Time Frame: Week 4
Measure: Count of Participants; unit: Participants
Arm/Group | Instruction Only | LHE-led
Number analyzed (Participants) | 109 | 104
Participants | 62 | 83

4. Secondary Outcome: Intention to Get Tested for COVID-19
Description: as for outcome 3
Time Frame: Week 8
Measure: Count of Participants; unit: Participants
Arm/Group | Instruction Only | LHE-led
Number analyzed (Participants) | 105 | 102
Participants | 70 | 82

ADVERSE EVENTS:
Time Frame: 8 weeks
Arm/Group | Instruction Only | LHE-led
All-Cause Mortality (participants affected / at risk) | 0/106 | 0/102
Serious Adverse Events (participants affected / at risk) | 0/106 | 0/102
Other Adverse Events (participants affected / at risk) | 0/106 | 0/102

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2022-11-16): https://cdn.clinicaltrials.gov/large-docs/82/NCT05435482/Prot_SAP_000.pdf